CLINICAL TRIAL: NCT04686539
Title: Synthetic CBD Oil Droplets as a Therapy for Mild to Moderate SARS-CoV-2 Infection. Assesment of Efficacy and Safety.
Brief Title: Synthetic CBD as a Therapy for COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Howard Amital, Head of Autoimmune Center, Head of internal medicine ward "B", Sheba Medical Center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-20-7526-HA-CTIL
Record Dates: First submitted 2020-12-18; First posted 2020-12-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Covid19; CBD
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recipients of CBD oil (Experimental): Patients receiving Cannabidiol oil drops, administered sublingual, 3 times a day, while hospitalized. Dosing and administration frequency would be assessed bi-daily by the medical staff.
  Interventions: Drug: CBD
- Recipients of Placebo (Placebo Comparator): Patients receiving placebo oil, administered sublingual, 3 times a day, while hospitalized.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD — CBD oil not containing THC, to be administered sub-lingual.
  Arms: Recipients of CBD oil
Drug: Placebo — Placebo Oil
  Arms: Recipients of Placebo

SUMMARY:
The study aim to test proof of concept of CBD treatment for efficacy and safety in patients suffering with mild COVID-19 infection. The CBD will be delivered via oil droplets not containing THC, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 patients
* 18 Years and older

Exclusion Criteria:

* Respiratory failure requiring mechanical ventilation
* Intensive care unit admission
* Neutrophile con. < 1000 cells/mm3
* Lymphocyte con < 500 cells/mm3
* Liver enzymes 5 times higher then the norm
* QT interval longer then 500 ms.
* Pregnancy
* Hemodialysis renal replacement therapy
* Active or prior psychotic event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Clinical deterioration | 14 days
  Patients chance of clinical deterioration of COVID19 disease as defined by percentage of patients requiring oxygen therapy during their hospitalization.

SECONDARY OUTCOMES:
Changes in NEWS scale | 14 days
  NEWS2- National Early Warning Score - a score defining the probability of severe COVID 19 disease. Minimum score is 0, while maximum score is 23. Higher score means worse outcome
Supportive care therapies | 14 days
  Percentage of patients requiring the respiratory support of either of the following : high flow nasal canula oxygen support, mechanical ventilation or use of extra corporeal membrane oxygenation.
SARS-COV2 presence | 10 days, 14 days
  Presence of SARS-COV2 in oral & nasal secretions in days 10, 14 of the study
Hospitalization Days | 14 days
  Hospitalization days due to COVID-19
Cytokine Levels | Day 3, day 7, discharge day (which is on average the 10th day of hospitalization).
  IL2, IL18, IL8. IL6, IL10, TNF-alpha, TGF-beta levels at day 3, day 7 and discharge day (which is on average the 10th day of hospitalization).
  All cytokine levels would be measured by pg/mL.
Hamilton Anxiety Score | 14 days
  A verified score measuring anxiety. Minimum score is 0, while maximum score is 56. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Amital, MD, MHA, Principal Investigator — Head of Internal Medicine ward "B", Sheba Health Center, Tel Hashomer
Locations (1):
- Sheba Medical Center, Tel Hashomer, Ramat Gan, Tel Aviv, Israel